CLINICAL TRIAL: NCT04388033
Title: Clinical Study of an Dendritic and Glioma Cells Fusion Vaccine With IL-12 for Treatment-naïve GBM Patients.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Medical Biotechnology Co., Ltd (Unknown); CyTIX.Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDKZJU-DCf12-2019408
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-12

CONDITIONS: Glioblastoma; Glioma; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms; Neoplasms, Nerve Tissue; Vaccines; Immunologic Factors
MeSH Terms: conditions — Glioblastoma; Glioma; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms; Neoplasms, Nerve Tissue | interventions — Interleukin-12; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety Evaluation Group (Experimental): Basic treatment phase:
  The patients have surgery followed by concomitant radiation (2 Gy/day x 30 days) and TMZ-chemotherapy (75 mg/m2/ day x 42 days).
  Immunotherapy phase:
  Maintenance chemotherapy with TMZ will be administered at 150-200 mg/m2/day for 5 days in each 28-day cycle. Fusion cells will be suspended in 0.5 mL normal saline and then injected intradermally close to a cervical lymph node. IL-12 will be injected subcutaneously at the same side at dose of 6ug twice for interval of one hour.
  Interventions: Biological: Dendritic Cell/Tumor Fusion Vaccine; Drug: Interleukin-12; Drug: Temozolomide

INTERVENTIONS:
Biological: Dendritic Cell/Tumor Fusion Vaccine — Vaccine is derived from the participants dendritic cells and tumor cells.
  Other Names: DC/tumor cell fusion vaccine
Drug: Interleukin-12 — Given subcutaneously at dose of 6ug twice for interval of one hour.
  Other Names: IL-12
Drug: Temozolomide — Following concomitant radiation (2 Gy/day x 30 days) and TMZ-chemotherapy (75 mg/m2/ day x 42 days) , maintenance chemotherapy with TMZ will be administered at 150-200 mg/m2/day for 5 days in each 28-day cycle.
  Other Names: TMZ

SUMMARY:
A multi-center, open-label, single-arm, phase I/II clinical study is designed to test the safety and immunogenicity of an investigational Dendritic and Glioma Cells Fusion vaccine given with IL-12 for treatment-naïve patients after resection of glioblastoma.

DETAILED DESCRIPTION:
This clinical trail includes two phases: basic treatment phase and immunotherapy phase. In basic treatment phase, patients will receive concomitant radiation and TMZ-chemotherapy. In immunotherapy phase, besides maintenance chemotherapy with TMZ, Fusion cells will be administered with IL-12 to enhance the immunity of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; Male or Female.
2. Treatment-naïve patients after Resection of Glioblastoma.
3. Histologically confirmed Glioblastoma.
4. KPS ≥ 60
5. White blood cell count (WBC) ≥ 3.0 x 109/L; peripheral blood lymphocyte (PBL) ≥ 25%.
6. Echocardiographic assessment of left ventricular ejection fraction (LVEF) ≥ 40% within 1 month of enrollment.
7. Patients must be able to understand the investigational nature of the study and provide informed consent.

Exclusion Criteria:

1. Those who are allergic constitution, or allergic to biological products, or have contraindications to CT and MRI1 contrast agents.
2. Those with severe autoimmune diseases or immunodeficiency diseases.
3. Those who are expected to take systemic corticosteroids within three months.
4. Those who needs long-term usage of immunosuppressive agents.
5. Those with infectious diseases, including syphilis, AIDS, hepatitis B, hepatitis C, etc.
6. Those who plan to receive any other anti-tumor treatment during the trial.
7. Combined with serious primary diseases of cardiovascular, liver and kidney, and liver function (ALT, AST, Y-GT) exceeding 1.5 times of the upper limit: BUN or Cr exceeding 1.5 times of the upper limit of normal value.
8. Patients with other malignant tumors.
9. Those with active infections, etc.
10. Suspected or confirmed a history of alcohol and drug abuse.
11. Psychiatric illness, intellectual and language disabilities that compromise the informed consent process, at the discretion of the investigator.
12. Women who are pregnant or nursing.
13. Women of childbearing age who refuse to contraception.
14. Active participation in another clinical treatment trials.
15. According to the judgment of the investigator, other conditions that the plan cannot be followed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) / Serious Adverse Events (SAE) | 2-3 years
  AE/SAE associated with the intervention will be captured throughout the treatment portion of the study. All adverse events will be then compiled and these patients will be recorded.
Progression free survival (PFS) at 6 months | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Assessed from this study start date to the date of the first observation of clinical or radiographic disease progression or death due to any cause. Patients will be censored at the time they are last known to be alive and progression free (if withdrawn or lost to follow-up).

SECONDARY OUTCOMES:
Immunological Assays | 2-3 years
  Assays including Flow Cytometry and Elispot will be employed to determine if cellular and humoral immunity were induced by serial vaccination with DC/Tumor Fusion Cells and IL-12.
Overall survival (OS) time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Assessed from this study start date to date of death of any cause. Patients will be censored at the time that they are last known to be alive (if withdrawn or lost to follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Shen, MD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No